CLINICAL TRIAL: NCT01902550
Title: A Randomized, Double-Blind, 2-Period Crossover Study to Evaluate the Effect of Single Dose JNJ-54452840 on Pharmacodynamics of Metoprolol Tartrate Immediate-Release in Healthy Subjects
Brief Title: A Crossover Study to Evaluate the Effect of JNJ-54452840 on Pharmacodynamics of Metoprolol Tartrate Immediate-Release in Healthy Participants
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Trial was stopped because study not required for development.
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CR102301; 54452840HFA1002
Record Dates: First submitted 2013-07-15; First posted 2013-07-18 (Estimated); Last update posted 2016-11-01 (Estimated); Status verified 2016-10

CONDITIONS: Healthy
Keywords: Healthy; JNJ-54452840; Metoprolol Tartrate Immediate-Release; Placebo; Male
MeSH Terms: interventions — JNJ-54452840

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Metoprolol plus placebo then Metoprolol plus JNJ-54452840 (Experimental): Metoprolol tartrate immediate-release (metoprolol IR) will be administered as single oral dose of 100 milligram (mg) tablet or capsule. After two hours, placebo (normal saline) will be administered intravenously over 1 minute on Day 1.
  Interventions: Drug: Metoprolol tartrate immediate-release (metoprolol IR); Drug: JNJ-54452840; Drug: Placebo
- Metoprolol plus JNJ-54452840 then Metoprolol plus placebo (Experimental): Metoprolol IR will be administered as single oral dose of 100 mg tablet or capsule. After two hours, JNJ-54452840 (12 milliliter [ml] solution containing 240 mg JNJ-54452840) will be administered intravenously over 1 minute.
  Interventions: Drug: Metoprolol tartrate immediate-release (metoprolol IR); Drug: JNJ-54452840; Drug: Placebo

INTERVENTIONS:
Drug: Metoprolol tartrate immediate-release (metoprolol IR) — Metoprolol IR will be administered as single oral dose of 100 mg tablet or capsule.
Drug: JNJ-54452840 — JNJ-54452840 (12 ml solution containing 240 mg JNJ-54452840) will be administered intravenously over 1 minute.
Drug: Placebo — Matching Placebo (normal saline) to JNJ-54452840 will be administered intravenously over 1 minute on Day 1.

SUMMARY:
The purpose of this study is to evaluate effect of co-administration of JNJ-54452840 and metoprolol tartrate immediate-release (metoprolol IR) compared to metoprolol IR alone on the exercise heart rate and blood pressure measured at the end of each 3-minute exercise test in healthy participants.

DETAILED DESCRIPTION:
This is a Phase 1, randomized (the study drug is assigned by chance), single-center, double-blind (neither physician nor participant knows the treatment that the participant receives) and 2-period crossover (participants may receive different interventions sequentially during the trial) study of JNJ-54452840 and metoprolol tartrate in healthy participants. The duration of study will be up to 7 weeks per participant and up to 1 year for participants if they develop anti-beta 1-AR (adrenergic receptor) auto-antibodies (auto-antibodies targeting the human beta-1-AR, antibody is a type of protein that helps protect the body against foreign matter, such as bacteria and viruses). The study consists of 3 parts: Screening (that is, up to 14 days before study commences on Day 1); Treatment (consists of either metoprolol IR and JNJ-54452840 or metoprolol IR and Placebo for 8 days, in subsequent two-treatment periods, separated by wash-out period of 2-7 days); and Follow-up (that is, 7-10 days after last study dose for safety assessment; followed by another visit after 21-28 days of last study dose for assessment of anti beta-1-AR auto-antibodies in blood). Any potential interaction between JNJ-54452840 and metoprolol tartrate IR will primarily be evaluated by measuring exercise induced heart rate (that is, post exercise). Participants' safety will be monitored throughout the study. If beta-1-AR-auto-antibodies are detected at the follow up visit 21-28 days after last treatment period study procedure, additional testing will be performed every 3 months until auto-antibody levels fall below the level of detection of the assay or for 1 year, whichever occurs earlier.

ELIGIBILITY:
Inclusion Criteria:

* Be a healthy non-smoking male with no clinically relevant abnormalities
* Able to perform upright bicycle ergometer exercise test and be able to achieve greater than or equal to 80 percent of maximum heart rate (HR) determined as (220 beats per minute [bpm]-age) during the last 10 seconds of the 3rd minute of exercise test
* Agree to abstain from caffeine (example, coffee, tea, chocolate, or caffeine-containing soft drinks) intake during the inpatient portion of the study
* Participants with body mass index between 18 and 32 kilogram per square meter (kg/m^2) and body weight greater than or equal to 50 kilogram (Kg) at screening

Exclusion Criteria:

* Contraindication to metoprolol tartrate immediate release (metoprolol IR)
* Resting HR less than 50 bpm and blood pressure less than 110/70 millimeter of mercury (mmHg)
* Physical disability that would preclude safe and adequate exercise test performance
* History of or current clinically significant medical illness that the Investigator considers should exclude the subject or that could interfere with the interpretation of the study results
* Determined to have variant cytochrome P4502D6 (CYP2D6) alleles encoding for altered metabolism
* Have a known or suspected intolerance or hypersensitivity to any biologic medication or known allergies or clinically significant reactions to murine, chimeric, or human peptides or proteins

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2013-07; Primary Completion 2013-10 (Estimated); Study Completion 2014-05 (Estimated)

PRIMARY OUTCOMES:
Exercise Heart Rate | Day 1 of Treatment Period 1
  Heart rate will be measured during the last 10 seconds of each 3-minute upright bicycle ergometer exercise test in healthy participants.
Exercise Heart Rate | Day 1 of Treatment Period 2
  Heart rate will be measured during the last 10 seconds of each 3-minute upright bicycle ergometer exercise test in healthy participants.

SECONDARY OUTCOMES:
Exercise Blood Pressure | Day 1 of Treatment Period 1 and 2
  Blood Pressure will be measured during the last 10 seconds of each 3-minute upright bicycle ergometer exercise test in healthy participants.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- Knoxville, Tennessee, United States